CLINICAL TRIAL: NCT05292040
Title: An Adaptive Design, Phase 1, Open-label Study to Investigate Receptor Occupancy in Brain After Single Oral Doses of LY3857210 as Measured by Positron Emission Tomography (PET) With the Radioligand [18F]-LY3818850 in Healthy Participants
Brief Title: A Study of LY3857210 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18313; J3O-MC-LSBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY3857210 (Experimental): Single doses of LY3857210 administered orally.
  Interventions: Drug: LY3857210

INTERVENTIONS:
Drug: LY3857210 — Administered orally.

SUMMARY:
The main purpose of this study is to evaluate the presence of study drug LY3857210 in the brain measured by positron emission tomography (PET) with the radioligand [18F]-LY3818850 in healthy participants. The safety and tolerability of LY3857210 will also be evaluated. The study will last up to approximately 6 weeks for each participant and may include up to four visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy male or female participants as determined by medical evaluation
* Have body weight ≥ 45 kilograms (kg) and body mass index (BMI) within the range 18.5 to 32.0 kilograms per square meter (kg/m²) (inclusive)
* Are males and in agreement to follow contraceptive requirements, or women of non-child-bearing potential

Exclusion Criteria:

* Have contraindications to undergoing magnetic resonance imaging (MRI) examination including but not limited to implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips, and other medical implants that have not been certified for head MRI
* Have clinically significant findings on the screening MRI scan, as judged by the investigator
* Suffer from claustrophobia and would be unable to tolerate the confined spaces of MRI or PET camera

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in brain receptor occupancy (RO) of LY3857210 measured by [18F]-LY3818850 PET scan | Baseline through study completion, up to approximately 6 weeks
  Change from baseline in brain RO of LY3857210 measured by [18F]-LY3818850 PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Invicro, Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No